CLINICAL TRIAL: NCT04561466
Title: Study of Efficacy of Befizal® 200 mg for the Treatment of Leber Hereditary Optic Neuropathy
Brief Title: Trial of Befizal® 200 mg for the Treatment of Leber Hereditary Optic Neuropathy
Acronym: Béfinohl
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hôpital Necker-Enfants Malades (Other)
Collaborators: European Georges Pompidou Hospital (Other); CLAIROP (Unknown)
Responsible Party: Principal Investigator, Christophe Orssaud, Principal investigator, Hôpital Necker-Enfants Malades
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: beza16
Record Dates: First submitted 2019-03-14; First posted 2020-09-23 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Safety Issues; Efficacy, Self
Keywords: leber herediatry optic neuropathy; befizal
MeSH Terms: interventions — Bezafibrate

STUDY DESIGN:
Intervention Model Description: open
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): 14 adult patients in whom the diagnosis of LHON obtained on anamnestic, clinical and ancillary testing / laboratory data. LHON should have occurred for less than 5 years and must be genetically proved with a 3460 or 11778 mitochondrial DNA mutation. Given the mode of transmission, genetic research may have been carried out in a maternal relative.
  Befizal® 200 mg will be tested for one year
  Interventions: Drug: Béfizal

INTERVENTIONS:
Drug: Béfizal — 600 mf befizal a day for one year

SUMMARY:
Study of the efficiency of Béfizal® 200 mg in 14 adult patients with a LHON that occurred for less than 5 years. Patient must have certain specific mutations

DETAILED DESCRIPTION:
Study of the efficiency of Béfizal® 200 mg in 14 adult patients in whom the diagnosis of LHON obtained on anamnestic, clinical and ancillary testing / laboratory data. LHON should have occurred for less than 5 years and must be genetically proved with a 3460 or 11778 mitochondrial DNA mutation. Given the mode of transmission, genetic research may have been carried out in a maternal relative

ELIGIBILITY:
Inclusion Criteria:

* Adult patients in whom the diagnosis of LHON obtained on anamnestic, clinical and ancillary testing / laboratory data. LHON should have occurred for less than 5 years and must be genetically proved with a 3460 or 11778 mitochondrial DNA mutation. Given the mode of transmission, genetic research may have been carried out in a maternal relative

Exclusion Criteria:

* * Any optic neuropathy for which the diagnosis of LHON is not formally confirmed or genetically proven;

  * LHON that started for more than 5 years;
  * LHON associated with another primary mutation than 3460 or 11778
  * Children or adult patients under guardianship or deprived of liberty by administrative or judicial decision;
  * Women of childbearing age ; pregnant or lactating women;
  * Patients who do not have affiliation to a social protection scheme (national or private insurance / beneficiary or assignee);
  * Patient who did not give its written, informed and signed consent;
  * Allergy to fibrate, bezafibrate and / or BEFIZAL® 200mg (Arrow Generiques) or one of these constituents;
  * Photosensitivity reactions related to fibrates;
  * Patient already receiving treatment with fibrates or HMG Co-A reductase inhibitors or anticoagulants;
  * Hepatic insuffisiency or dysfunction with increased of transaminases (AST and ALT) over 3 times of the normal;
  * Renal insufficiency with serum creatinine> 15 mg / L (> 135 mg / dL) Biliary pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Evolution of best corrected farsight visual acuity (in LogMAR) | Month12
  Measurement of the best corrected farsight visual acuity by Early Treatment Diabetic Retinopathy Study type scale (range from -0.3 to 2.6) -0.3 is the best vision and 2.6 the worse

SECONDARY OUTCOMES:
Farsight best corrected visual acuity | Month 3
  Measurement of the Farsight best corrected visual acuity in LogMAR by Early Treatment Diabetic Retinopathy Study type scale (range from -0.3 to 2.6) -0.3 is the best vision and 2.6 the worse
Evolution of Farsight best corrected visual acuity | Month 6
  Measurement of the Farsight best corrected visual acuity in LogMAR by Early Treatment Diabetic Retinopathy Study type scale (range from -0.3 to 2.6) -0.3 is the best vision and 2.6 the worse
Evolution of Farsight best corrected visual acuity | Month 9
  Measurement of the Farsight best corrected visual acuity in LogMAR by Early Treatment Diabetic Retinopathy Study type scale (range from -0.3 to 2.6) -0.3 is the best vision and 2.6 the worse
Evolution of Farsight best corrected visual acuity | Month 15
  Measurement of the Farsight best corrected visual acuity in LogMAR by Early Treatment Diabetic Retinopathy Study type scale (range from -0.3 to 2.6) -0.3 is the best vision and 2.6 the worse
Evolution of Farsight best corrected visual acuity | Month 3
  Measurement of the Farsight best corrected visual acuity by Early Treatment Diabetic Retinopathy Study type scale (range from -0.3 to 2.6) -0.3 is the best vision and 2.6 the worse
Evolution of Farsight decimal best corrected visual acuity | Month 6
  Measurement of the Farsight best corrected visual acuity (in LogMAR) measured with a Monoyer scale (range from 20/20 to light perception). 20/20 is the best vision and light perception the worse
Evolution of Farsight decimal best corrected visual acuity | Month 9
  Measurement of the Farsight best corrected visual acuity (in LogMAR) measured with a Monoyer scale (range from 20/20 to light perception). 20/20 is the best vision and light perception the worse
Evolution of Farsight decimal best corrected visual acuity | Month 12
  Measurement of the Farsight best corrected visual acuity (in LogMAR) measured with a Monoyer scale (range from 20/20 to light perception). 20/20 is the best vision and light perception the worse
Evolution of Farsight decimal best corrected visual acuity | Month 15
  Measurement of the Farsight best corrected visual acuity (in LogMAR) measured with a Monoyer scale (range from 20/20 to light perception). 20/20 is the best vision and light perception the worse
Evolution of Nearsight visual acuity | Month 3
  Measurement of the best corrected nearsight visual acuity measured using a Parinaud scale (from P48 to P1>.5) P48 is the worse vision and P1.5 the best
Evolution of Nearsight visual acuity | Month 6
  Measurement of the best corrected nearsight visual acuity measured using a Parinaud scale (from P48 to P1>.5) P48 is the worse vision and P1.5 the best
Evolution of Nearsight visual acuity | Month 9
  Measurement of the best corrected nearsight visual acuity measured using a Parinaud scale (from P48 to P1>.5)P48 is the worse vision and P1.5 the best
Evolution of Nearsight visual acuity | Month 12
  Measurement of the best corrected nearsight visual acuity measured using a Parinaud scale (from P48 to P1>.5) P48 is the worse vision and P1.5 the best
Evolution of Nearsight visual acuity | Month 15
  Measurement of the best corrected nearsight visual acuity measured using a Parinaud scale (from P48 to P1>.5) P48 is the worse vision and P1.5 the best
Evolution of retinal nerve fibers layer Optical Coherent Tomography | Month 6
  physiological parameter : Optical Coherent Tomography
Evolution of retinal nerve fibers layer Optical Coherent Tomography | Month 12
  physiological parameter : Optical Coherent Tomography
automated visual field measurement | Month 3
  physiological parameter : automated visual field corrected deviation of a visual field, measured according to a protocol STAT protocol 30 (Champ visuel Métrovision, Perenchies, France)
automated visual field measurement | Month 6
  physiological parameter : automated visual field
automated visual field | Month 9 of a treatment with BEFIZAL® 200mg (ARROW GENERIQUES) compare to Month 0
  physiological parameter : automated visual field corrected deviation of a visual field, measured according to a protocol STAT protocol 30 (Champ visuel Métrovision, Perenchies, France)
automated visual field measurement | Month 12
  physiological parameter : automated visual field corrected deviation of a visual field, measured according to a protocol STAT protocol 30 (Champ visuel Métrovision, Perenchies, France)
automated visual field measurement | Month 15
  physiological parameter : automated visual field corrected deviation of a visual field, measured according to a protocol STAT protocol 30 (Champ visuel Métrovision, Perenchies, France)
Manual visual field measurement | Month 3
  physiological parameter : manual visual field measured with isopters V / 4, III / 1 and II / 1
Manual visual field measurement | Month 6
  physiological parameter : manual visual field measured with isopters V / 4, III / 1 and II / 1
Manual visual field measurement | Month 9
  physiological parameter : manual visual field measured with isopters V / 4, III / 1 and II / 1
Manual visual field measurement | Month 12
  physiological parameter : manual visual field measured with isopters V / 4, III / 1 and II / 1
Manual visual field measurement | Month 15
  physiological parameter : manual visual field measured with isopters V / 4, III / 1 and II / 1
National Eye Institute Visual Function Questionnaire 25 | Month 12
  Questionnaire
Concentration of serum creatinine | Every three months until Month 15
  Concentration of serum creatinine
Concentration of high-density lipoprotein cholesterol | Every three months until Month 15
  Blood test
Concentration of very low-density lipoprotein cholesterol | Every three months until Month 15
  Blood test
Concentration of triglycerides | Every three months until Month 15
  Blood test
Rate of Partial thromboplastin time | Every three months until Month 15
  Blood test
Concentration of Aspartate aminotransférase | Every three months until Month 15
  Blood test
Concentration of Alanine aminotransférase | Every three months until Month 15
  Blood test
Concentration of lactate deshydrogenase | Every three months until Month 15
  Blood test
Concentration of creatine kinase | Every three months until Month 15
  Blood test

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Bremond Gignac, MD PhD, Study Chair — Necker Hopsital
Locations (1):
- HEGP Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided
Undecided